CLINICAL TRIAL: NCT06034899
Title: A Phase 1, 2-part, Open-label, Randomized, 2-period, 2-sequence, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of BMS-986196 Phase 2 Tablet Formulation at Two Dose Levels in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effect of Food on the Drug Levels of BMS-986196 in Healthy Adult Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM038-1014
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Adult Volunteers
Keywords: BMS-986196; Healthy adult participants; Pharmacokinetics; Cross-over study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: BMS-986196 Dose 1 (Treatment A) (Experimental)
  Interventions: Drug: BMS-986196
- Part 1: BMS-986196 Dose 1 (Treatment B) (Experimental)
  Interventions: Drug: BMS-986196
- Part 2: BMS-986196 Dose 2 (Treatment A) (Experimental)
  Interventions: Drug: BMS-986196
- Part 2: BMS-986196 Dose 2 (Treatment B) (Experimental)
  Interventions: Drug: BMS-986196

INTERVENTIONS:
Drug: BMS-986196 — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the drug levels of BMS-986196 and to evaluate the effect of food (fasted versus fed [high-fat meal]) on the drug levels after administration of BMS-986196 tablet formulation at two dose levels in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants and female participants without clinically significant deviation from normal, as determined by the investigator, in medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory assessments.
* Body mass index of 18.0 to 35.0 kilograms/meter square (kg/m^2), inclusive, and body weight ≥ 50 kg.
* Participant must agree and be willing to consume a standard high-fat meal (for example, which may contain gluten).

Exclusion Criteria:

* Any significant acute or chronic medical illness in the assessment of the investigator.
* Current or recent (within 3 months of study intervention) gastrointestinal (GI) disease that could possibly affect drug absorption, distribution, metabolism, and excretion (e.g., bariatric procedure)
* Any major surgery, including GI surgery (for example, cholecystectomy and any other GI surgery) that could impact upon the absorption of study intervention (uncomplicated appendectomy and hernia repair are acceptable).

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-22 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Predose and post-dose up to Day 10
Maximum observed serum concentration (Cmax) | Predose and post-dose up to Day 10
Time of Cmax (Tmax) | Predose and post-dose up to Day 10

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to Day 36
Number of participants with serious AEs (SAEs) | Up to Day 36
Number of participants with vital sign abnormalities | Up to Day 11
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 11
Change from baseline in columbia-suicide severity rating scale (C-SSRS) at day 11 | Baseline, Day 11
Number of participants with physical examination findings | Up to Day 11
Number of participants with clinical laboratory abnormalities | Up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com